CLINICAL TRIAL: NCT05537974
Title: Effect of Endotracheal Aspiration on End-expiratory Lung Volume in Patients With ARDS, Comparison of Open vs. Closed Suction, A Randomize Cross-over Study
Brief Title: Open Suction vs. Closed Suction in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Professor Doctor, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IGHCEAH-ICU-7
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Endotracheal aspiration, Electric impedance tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This is a crossover study and suction procedure was made in a random order with 60 minutes wash out period between two suction maneuvers. Patients were randomized after intubation; randomization was made with sealed envelopes.
  All patients mechanically ventilated with lung protective ventilation strategy. Before the suctioning the patients ventilated with 100% of oxygen for 60 seconds. In open suction, the patient was disconnected from mechanical ventilator, the aspiration catheter advanced until resistance met after that the catheter withdraw 1 cm before aspiration. During endotracheal suctioning a negative pressure applied two times for 5 seconds. The negative pressure was set 150 mmHg. All suctioning maneuvers performed by intensivists.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Suction (Other): Endotracheal aspiration will perform after the patient disconnect from mechanical ventilation
  Interventions: Procedure: Endotracheal aspiration
- Closed Suction (Other): Endotracheal aspiration will perform without disconnection from mechanical ventilation
  Interventions: Procedure: Endotracheal aspiration

INTERVENTIONS:
Procedure: Endotracheal aspiration — Clearance of endotracheal secretions via a catheter.

SUMMARY:
The alveoli tend to collapse in patients with ARDS. Endotracheal aspiration may increase alveolar collapse by decreasing the end-expiratory lung volume. The hypothesis is that closed endotracheal aspiration led to less end-expiratory volume loss when compared to open endotracheal aspiration.

ELIGIBILITY:
Inclusion Criteria:

Mechanically ventilated due to ARDS

Exclusion Criteria:

Hemodynamically unstable Air leaks syndrome (pneumothorax) Higher level of FiO2 (>60%) Chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
End expiratory lung volume (EELV) | One minute before suctioning, 1, 10, 20, 30 minutes after suctioning
  End expiratory lung impedance (EELI) will be measured wit electric impedance tomography. Change in EELI representative of change in EELV.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Dr Suat Seren Chest Diseases and Chest Surgery Training and Research Hospital, Intensive Care Unit, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildirim S, Saygili SM, Sunecli O, Kirakli C. Comparison of the effects of open and closed aspiration on end-expiratory lung volume in acute respiratory distress syndrome. Korean J Anesthesiol. 2024 Feb;77(1):115-121. doi: 10.4097/kja.23194. Epub 2023 May 22. PMID 37211764